CLINICAL TRIAL: NCT01950858
Title: Safety and Efficacy of Hyper Baric Oxygen Therapy (HBOT) in Patients Presenting With Spontaneous Osteonecrosis of the Knee
Brief Title: Hyper Baric Oxygen Therapy (HBOT) for Spontaneous Osteonecrosis of the Knee
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Yiftah Beer, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91/12*1
Record Dates: First submitted 2013-08-28; First posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Spontaneous Osteonecrosis of the Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biological (Experimental): 6 weeks of HBO treatment as well as non weight bearing
  Interventions: Biological: Weight reduction
- Control (Active Comparator): non weight bearing
  Interventions: Biological: Weight reduction

INTERVENTIONS:
Biological: Weight reduction

SUMMARY:
safety and efficacy of Hyper Baric Oxygen (HBO) in patients presenting with spontaneous osteonecrosis of the knee

ELIGIBILITY:
Inclusion Criteria:

* Age40-85 years
* Diagnosis of Spontaneous osteonecrosis of the knee (SONK)in last month, Stage 1 or 2 by MRI.

Exclusion Criteria:

* Hyperbaric treatment (HBOT) in the last 2 years.
* Any contraindication for HBOT
* Pregnancy.
* Inability to sign inform consent
* Any contraindication for MRI

Ages: 40 Months to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 6 weeks
  Pain Reduction
Safety | end of HBOT
  Number of Participants with Adverse Events during HBOT

SECONDARY OUTCOMES:
Reduction In AVN size by MRI | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel